CLINICAL TRIAL: NCT02727439
Title: Influence of Acute Exhausting Exercise on Microvascular Reactivity in Healthy Sedentary Subjects and Athletes
Brief Title: Acute Exercise and Microvascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Ines Drenjancevic, Vice Dean for Science, Faculty of Medicine Josip Juraj Strossmayer University of Osijek, Josip Juraj Strossmayer University of Osijek
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 215861071403
Record Dates: First submitted 2016-03-18; First posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Physical Exertion
Keywords: microvascular function; laser Doppler flowmetry; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sedentary Subjects (Experimental): Healthy lean sedentary subjects.
  Interventions: Other: Acute Exhausting Exercise (AE)
- Athletes (Experimental): Active athletes.
  Interventions: Other: Acute Exhausting Exercise (AE)

INTERVENTIONS:
Other: Acute Exhausting Exercise (AE) — A single progressive rowing training to maximal exhaustion (AE).

SUMMARY:
It is well recognized that chronic exercise protects against the development of cardiovascular diseases. However, the responses of vasculature to acute exercise (AE) are not well known and not consistent in literature. Acute exertional exercise can induce large, transient increases in arterial pressure and development of metabolic acidosis which can be associated with pro-inflammatory response involving oxidant stress and circulating cytokines known to impair endothelial function.

The aim of this study is to test the impact of a single exposure to exhausting training on microvascular reactivity in healthy sedentary subjects and athletes.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* active athletes
* lean sedentary subjects

Exclusion Criteria:

* drugs that could affect the endothelium
* overweight
* hypertension
* coronary artery disease
* diabetes
* hyperlipidaemia
* renal impairment
* cerebrovascular and peripheral artery disease

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Skin microcirculation post occlusive reactive hyperemia | Post occlusive reactive hyperemia - PORH, recorded by Laser Doppler Flowmetry will be measured immediately after acute exhausting training.
  Cutaneous microvascular blood flow will be measured by Laser Doppler Flowmetry in response to vascular occlusion (post occlusive reactive hyperemia - PORH) before and after acute exhausting training.
Skin microcirculation acetylcholine induced dilation | Acetylcholine induced dilation (AChID), recorded by Laser Doppler Flowmetry will be measured immediately after acute exhausting training.
  Cutaneous microvascular blood flow will be measured by Laser Doppler Flowmetry in response to iontophoresis of acetylcholine (acetylcholine induced dilation, AChID) before and after acute exhausting training.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Drenjancevic, MD, PhD, Principal Investigator — Faculty of Medicine, Josip Juraj Strossmayer University of Osijek
Locations (1):
- Faculty of Medicine Osijek, Laboratory for Clinical and Sport Physiology, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavka A, Cosic A, Jukic I, Jelakovic B, Lombard JH, Phillips SA, Seric V, Mihaljevic I, Drenjancevic I. The role of cyclo-oxygenase-1 in high-salt diet-induced microvascular dysfunction in humans. J Physiol. 2015 Dec 15;593(24):5313-24. doi: 10.1113/JP271631. Epub 2015 Dec 7. PMID 26498129
- [Background] Cavka A, Jukic I, Ali M, Goslawski M, Bian JT, Wang E, Drenjancevic I, Phillips SA. Short-term high salt intake reduces brachial artery and microvascular function in the absence of changes in blood pressure. J Hypertens. 2016 Apr;34(4):676-84. doi: 10.1097/HJH.0000000000000852. PMID 26848993
- [Background] Phillips SA, Das E, Wang J, Pritchard K, Gutterman DD. Resistance and aerobic exercise protects against acute endothelial impairment induced by a single exposure to hypertension during exertion. J Appl Physiol (1985). 2011 Apr;110(4):1013-20. doi: 10.1152/japplphysiol.00438.2010. Epub 2011 Jan 20. PMID 21252216